CLINICAL TRIAL: NCT00941109
Title: A Phase 1 Open-Label, Dose Escalation Study to Determine the Absolute Bioavailability of a Single Oral Dose Administration of Decitabine in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Escalation Study to Determine Bioavailability of a Single Oral Dose of Decitabine in Patients With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7373-A001-101
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: decitabine
- 2 (Experimental)
  Interventions: Drug: decitabine
- 3 (Experimental)
  Interventions: Drug: decitabine
- 4 (Experimental)
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine — Cohort 1: 30 mg oral on Day 1 and 20 mg/m^2 1-hour IV infusion on Days 2-5 of Cycle 1.
  Other Names: Dacogen
  Arms: 1
Drug: decitabine — Cohort 2: 60 mg oral on Day 1 and 20 mg/m^2 1-hour IV infusion on Days 2-5 of Cycle 1.
  Other Names: Dacogen
  Arms: 2
Drug: decitabine — Cohort 3: 120 mg oral on Day 1 and 20 mg/m^2 1-hour IV infusion on Days 2-5 of Cycle 1.
  Other Names: Dacogen
  Arms: 3
Drug: decitabine — Cohort 4: 240 mg oral on Day 1 and 20 mg/m^2 1-hour IV infusion on Days 2-5 of Cycle 1.
  Other Names: Dacogen
  Arms: 4

SUMMARY:
The purpose of this study is to determine how the body absorbs decitabine when taken orally in patients with Myelodysplastic Syndrome (MDS). Safety will also be assessed for this oral dose.

DETAILED DESCRIPTION:
Cohorts are dosed sequentially, and escalation may stop before the 5th cohort is dosed. Each cycle will be approximately 4 weeks in length. Following Cycle 1, patients may receive an additional 4 follow-up cycles of decitabine. Cycles 2-5 will include a 20 mg/m^2 1-hour IV infusion of decitabine on Days 1-5 for all cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed de novo or secondary MDS.
2. Age greater than or equal to 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
4. Adequate renal and hepatic function (creatinine less than or equal to 2.0 mg/dL, total bilirubin less than 2.0 mg/dL, aspartate aminotransferase [AST] or alanine aminotransferase [ALT] less than 3 times the upper limit of normal).
5. Life expectancy of at least 6 weeks.
6. If currently receiving 5 day decitabine regimen, patient must be scheduled to receive one more cycle of 5 day decitabine.
7. Recovered from all toxic effects of all prior therapy before entry into this study.
8. Women of childbearing potential and all men must agree to practice a medically approved form of contraception (one of the following must be used: condoms [male or female] with a spermicidal agent, diaphragm or cervical cap with a spermicidal agent, intrauterine device, hormonal contraception, abstinence) during the course of the study and up to 2 months following the last dose of decitabine.

Exclusion Criteria:

1. Candidates for up front high dose induction chemotherapy. MDS patients who are scheduled to receive decitabine prior to a bone marrow transplant or stem cell transplant are allowed.
2. History of treatment failure with decitabine.
3. Received any experimental agent within the preceding 30 days prior to screening.
4. Uncontrolled cardiac or pulmonary disease.
5. History of intestinal surgery, pancreatic surgery, or gastric surgery.
6. Any clinically relevant disease, disorder (including psychiatric disorders), or condition, in the opinion of the Investigator, which may interfere with the objectives of the study, especially with the gastrointestinal (GI) absorption of the study drug, and/or with the safety of the subject in the study.
7. Current active colitis of any etiology (Clostridium difficile colitis, ulcerative colitis, Crohn's disease, etc.) or a recent (less than 2 weeks) episode of colitis.
8. Pregnant or lactating. Female patients of childbearing potential must have had a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 prior to dosing.
9. Known positive serology for human immunodeficiency virus (HIV).
10. Active viral, fungal, or bacterial infection. No patient may enter the study unless infections have been fully treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) endpoints will be decitabine PK parameters: Tmax, Cmax, AUC0-inf, t1/2 and F. | Cycle 1 on Days 1 and 2 from predose up to 6 hours after administration.

SECONDARY OUTCOMES:
Safety evaluations will include assessments of adverse events (AEs), medical history, physical examinations, vital signs measurements, use of concomitant medications, and laboratory assessments at baseline and throughout the study period. | Up to 30 days after the last dose of decitabine

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Inc.
Locations (6):
- United States (6):
  - Scottsdale, Arizona
  - Denver, Colorado
  - Rochester, Minnesota
  - The Bronx, New York
  - Houston, Texas
  - Tacoma, Washington